CLINICAL TRIAL: NCT06697431
Title: A Randomized, Controlled, Open-label, Non Inferiority KawasakI Trial With Anakinra
Brief Title: Non Inferiority KawasakI Trial With Anakinra
Acronym: NIKITA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: Asst Degli Spedali Civili Di Brescia (Other); IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Gabriele Simonini, Professor, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIKITA
Record Dates: First submitted 2024-11-01; First posted 2024-11-20 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Kawasaki Disease; Anakinra
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein; Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Patients who fulfill the eligibility criteria and whose parent/carer (legal representative) have provided informed consent will be randomized 1:1 to receive standard of care IVIG and aspirin or anakinra and ASA.
  As epidemiological data suggest worse outcomes in terms of CAA for very young patients (age <1 years), in this setting, proper randomisation 1:1 procedure will be matched for age < or> than 1 year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anakinra (Experimental): Anakinra 2mg/kg intravenously, max 100 mg/dose 4 times/day
  Interventions: Drug: Anakinra
- Intravenous immunoglobulins (Active Comparator): IVIG 2g/kg administered in 10-12 hours as per local standard of care
  Interventions: Drug: Intravenous Immunoglobulins, Human

INTERVENTIONS:
Drug: Anakinra — Patients who fulfill the eligibility criteria a will be randomized 1:1 to receive either
  1. IVIG 2g/kg administered in 10-12 hours as per local standard of care (standard treatment) OR
  2. Anakinra 2mg/kg intravenously, max 100 mg/dose 4 times/day (investigational treatment)
  Patients showing fever, between 36 hours and 72 hours from the end of first line treatment will be considered failures. Failures from the investigational treatment arm will receive a dose of IVIG and they will drop from the study.
  Children who remained afebrile between the 36th and 72nd hour will be considered as responders, and they will proceed into the study.
  Patients in the standard treatment arm will continue ancillary treatment and follow-up .
  Patients in the investigational treatment arm will enter the tapering phase.
  Other Names: Kineret
  Arms: Anakinra
Drug: Intravenous Immunoglobulins, Human — see previous section
  Other Names: IVIG
  Arms: Intravenous immunoglobulins

SUMMARY:
This is a multicenter, open-label, randomized, controlled, interventional trial followed by a long-term observational extension period in patients with Kawasaki Disease (KD) to be treated eitherwith endovenous Immunoglobulins (IVIG-standard treatment) versus anakinra

Aim of the study: to demonstrate that anakinra is non-inferior to IVIG in KD, in terms of fever control in the acute phase and development of coronary artery dilation/aneurisms (CAA) within one year from the onset.

DETAILED DESCRIPTION:
This is a multicenter national, open label, randomized, controlled, interventional trial followed by a long-term observational extension period. This is a non-inferiority study Patients who fulfill the eligibility criteria and whose parent/carer (legal representative) has provided informed consent will be randomized 1:1 to receive either

1. IVIG 2g/kg administered in 10-12 hours as per local standard of care (standard treatment) OR
2. Anakinra 2mg/kg intravenously, max 100 mg/dose 4 times/day (investigational treatment)

PLUS Aspirin (ASA) 50mg/kg QID until 36 hours from fever disappearance, then switched to low-dose (3-5 mg/Kg once a day) as per standard of care

ELIGIBILITY:
Inclusion Criteria

1. KD defined in at least one of the three following ways as per American Heart Association (AHA) criteria: Fever for at least 5 days in addition to 4 of the following 5 clinical criteria:

   * bilateral non-purulent conjunctivitis
   * cervical lymphadenopathy
   * polymorphous skin rash
   * changes in lips or mucosa (strawberry tongue, red cracked lips, diffuse erythematous oropharynx)
   * extremity changes (erythema, oedema of palms and soles in initial phase, and at convalescent stage skin peeling)
2. less than 5 days of fever but all 5 clinical criteria above
3. incomplete KD cases defined as:

   * children/adolescents (>1 year old) with fever greater than or equal to 5 days AND at least 2 other compatible clinical criteria as listed above;
   * OR infants ≤ 1 year old with fever greater than or equal to 7 days without other explanation;

   AND for both age groups, CRP ≥30 mg/L or erythrocyte sedimentation rate (ESR) ≥40 mm/hr (or both) AND for both age groups EITHER the presence of any 3 or more of: anaemia for age (haemoglobin < lower limit of normal reference range for local laboratory); platelet count ≥450,000/L or <140,000/L; albumin <30 g/L; elevated ALT (> upper limit of normal reference range for local laboratory); white cell count ≥15,000/L; urine ≥10 white blood cells per high power field iv.

   OR abnormal echocardiogram compatible with KD but without established CAA, with ≥ 3 of the following suggestive features: decreased left ventricular function, mitral regurgitation, pericardial effusion, or dilated but non-aneurysmal coronary arteries (internal diameter 2≤Z<2.5; and not meeting the exclusion criteria for aneurysmal change as defined below).
4. To be enrolled children need to show persistent fever ≤7 days
5. Written informed consent from an appropriate legal representative(s), and assent from patients older than 7 years

Exclusion Criteria

1. Patients with KD and already established coronary artery aneurysms (CAA), as per AHA definition, at screening.
2. Clinical picture consistent with Kawasaki Shock Syndrome (KDSS) or Macrophage Activation Syndrome (MAS) OR Multisystem Inflammatory Syndrome in Children (MIS-C)
3. History or evidence of any previous heart disease
4. Known hypersensitivity to anakinra, IVIG and ASA or any medical condition that contraindicates the use of these treatments
5. Patients with KD receiving IVIG, corticosteroids, immunosuppressants, biologic treatments at the time of screening

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment response in both treatment arms | 12 months
  Response rate
Number of patients with CAA (as per Z-scores) at the end of the study period in both treatment arms | 12 months
  CAA rate in both arms. CAAs will be classified in accordance with the scheme based on Z scores proposed by AHA. No coronary involvement with Z score <2, dilation only with Z score > 2 to <2.5 or if initially <2 with a decrease during follow-up ≥1 3, small aneurysm with Z score ≥2.5 to <5, medium aneurysm with Z score ≥5 to <10 and absolute dimension <8 mm and large or giant aneurysm with Z score ≥10, or absolute dimension ≥8 mm

SECONDARY OUTCOMES:
Number of days with fever in both treatment arms | 90 days
  Fever as defined as T>38°C
Time to reach CRP values<50% from the highest value and to normalize it in both treatment arms (days) | 90 days
  CRP values expressed in mg/dL
Time to normalize coronary artery abnormalities (days) | 90 days
  CAAs will be classified in accordance with the scheme based on Z scores proposed by AHA. No coronary involvement with Z score <2, dilation only with Z score > 2 to <2.5 or if initially <2 with a decrease during follow-up ≥1 3, small aneurysm with Z score ≥2.5 to <5, medium aneurysm with Z score ≥5 to <10 and absolute dimension <8 mm and large or giant aneurysm with Z score ≥10, or absolute dimension ≥8 mm
Severity of coronary artery abnormalities (as per Z-score) at the end of follow-up | 24 months
  CAAs will be classified in accordance with the scheme based on Z scores proposed by AHA. No coronary involvement with Z score <2, dilation only with Z score > 2 to <2.5 or if initially <2 with a decrease during follow-up ≥1 3, small aneurysm with Z score ≥2.5 to <5, medium aneurysm with Z score ≥5 to <10 and absolute dimension <8 mm and large or giant aneurysm with Z score ≥10, or absolute dimension ≥8 mm
Length of hospitalization in both treatment arms (days) | 90 days
  Defined by days of hospitalization from disease onset to discharge
Time to stop anakinra (days) | 90 days
  From the first administration iv to the last sc
Adverse event and severe adverse event developed during the study and follow/up period | 24 months
  Medical Dictionary for Regulatory Activities (MeDRA) will be used for the description of adverse events (AEs), according to the regulatory requirements
Cumulative drug exposure (mg/kg/day) | 12 months
  Calculated for both iv e sc administration

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Simonini, Prof, Principal Investigator — Meyer Children's Hospital IRCCS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang J, Jain S, Capparelli EV, Best BM, Son MB, Baker A, Newburger JW, Franco A, Printz BF, He F, Shimizu C, Hoshino S, Bainto E, Moreno E, Pancheri J, Burns JC, Tremoulet AH. Anakinra Treatment in Patients with Acute Kawasaki Disease with Coronary Artery Aneurysms: A Phase I/IIa Trial. J Pediatr. 2022 Apr;243:173-180.e8. doi: 10.1016/j.jpeds.2021.12.035. Epub 2021 Dec 23. PMID 34953816
- [Background] Kone-Paut I, Tellier S, Belot A, Brochard K, Guitton C, Marie I, Meinzer U, Cherqaoui B, Galeotti C, Boukhedouni N, Agostini H, Arditi M, Lambert V, Piedvache C. Phase II Open Label Study of Anakinra in Intravenous Immunoglobulin-Resistant Kawasaki Disease. Arthritis Rheumatol. 2021 Jan;73(1):151-161. doi: 10.1002/art.41481. Epub 2020 Nov 17. PMID 32779863
- [Background] Kessel C, Kone-Paut I, Tellier S, Belot A, Masjosthusmann K, Wittkowski H, Fuehner S, Rossi-Semerano L, Dusser P, Marie I, Boukhedouni N, Agostini H, Piedvache C, Foell D. An Immunological Axis Involving Interleukin 1beta and Leucine-Rich-alpha2-Glycoprotein Reflects Therapeutic Response of Children with Kawasaki Disease: Implications from the KAWAKINRA Trial. J Clin Immunol. 2022 Aug;42(6):1330-1341. doi: 10.1007/s10875-022-01301-w. Epub 2022 Jun 14. PMID 35699824
- [Background] Blonz G, Lacroix S, Benbrik N, Warin-Fresse K, Masseau A, Trewick D, Hamidou M, Stephan JL, Neel A. Severe Late-Onset Kawasaki Disease Successfully Treated With Anakinra. J Clin Rheumatol. 2020 Mar;26(2):e42-e43. doi: 10.1097/RHU.0000000000000814. No abstract available. PMID 32073531
- [Background] Bossi G, Codazzi AC, Vinci F, Clerici E, Regalbuto C, Crapanzano C, Veraldi D, Moiraghi A, Marseglia GL. Efficacy of Anakinra on Multiple Coronary Arteries Aneurysms in an Infant with Recurrent Kawasaki Disease, Complicated by Macrophage Activation Syndrome. Children (Basel). 2022 May 5;9(5):672. doi: 10.3390/children9050672. PMID 35626849
- [Background] Maniscalco V, Abu-Rumeileh S, Mastrolia MV, Marrani E, Maccora I, Pagnini I, Simonini G. The off-label use of anakinra in pediatric systemic autoinflammatory diseases. Ther Adv Musculoskelet Dis. 2020 Oct 16;12:1759720X20959575. doi: 10.1177/1759720X20959575. eCollection 2020. PMID 33149772
- [Background] Gambacorta A, Buonsenso D, De Rosa G, Lazzareschi I, Gatto A, Brancato F, Pata D, Valentini P. Resolution of Giant Coronary Aneurisms in a Child With Refractory Kawasaki Disease Treated With Anakinra. Front Pediatr. 2020 May 7;8:195. doi: 10.3389/fped.2020.00195. eCollection 2020. PMID 32457855
- [Background] Mastrolia MV, Abbati G, Signorino C, Maccora I, Marrani E, Pagnini I, Simonini G. Early anti IL-1 treatment replaces steroids in refractory Kawasaki disease: clinical experience from two case reports. Ther Adv Musculoskelet Dis. 2021 Mar 29;13:1759720X211002593. doi: 10.1177/1759720X211002593. eCollection 2021. PMID 33854568